CLINICAL TRIAL: NCT02598687
Title: A Phase I Trial Testing TH-302, a Tumor-selective Hypoxia-Activated Cytotoxic Prodrug, in Combination With Preoperative Chemoradiotherapy in Patients With Distal Esophageal and Esophago-gastric Junction Adenocarcinoma
Brief Title: Testing TH-302, in Combination With Preoperative Chemoradiotherapy, in Esophageal Cancer.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 2 Phase 3 trials didn't meet their primary endpoint, so further development and testing of TH-302 is uncertain
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Threshold Pharmaceuticals (Industry); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-27-03/09
Record Dates: First submitted 2015-05-29; First posted 2015-11-06 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — TH 302; Carboplatin; Paclitaxel; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Other): treatment arm: TH-302 pre-treatment day 4 and weekly during treatment. 5 x carboplatin and paclitaxel, radiotherapy: 23 x 1.8Gy HX4 scans day 1 and day 8,surgery 6-10 weeks after chemo-radiotherapy
  Interventions: Drug: TH-302; Other: HX4 scan; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiotherapy; Procedure: surgery

INTERVENTIONS:
Drug: TH-302 — TH-302 day 4 (pre-treatment) and weekly during chemo-radiotherapy (CRT)
Other: HX4 scan — HX 4 scan day 1 and day 8
Drug: Carboplatin — 2mg/ml/min
Drug: Paclitaxel — 50 mg/m2
Radiation: Radiotherapy — 23 x 1.8 Gy
Procedure: surgery — minimally invasive transhiatal approach including a one-field node dissection or transthoracic approach with a two-field lymph node dissection

SUMMARY:
Open-label, single-center phase 1 study of an investigational agent TH-302 and standard chemoradiotherapy with a 3+3 dose escalation design through 3 dose levels.

DETAILED DESCRIPTION:
Rationale:

Neoadjuvant chemoradiotherapy followed by surgery remains the standard of care for esophageal cancer patients. Both limited local response as well as distant metastases are a common cause of treatment failure. Combining TH-302 with chemo-radiotherapy may improve outcome by:

* Direct cytotoxic effect of TH-302 on hypoxic cells of the primary tumor without enhancing normal tissue toxicity.
* Increase the sensitivity of the primary tumor to chemo-radiotherapy by decreasing the hypoxic fraction.
* A bystander cytotoxic effect of TH-302 on normoxic cells adjacent to hypoxic cells of the primary tumor.
* A potential cytotoxic effect on micro-metastasis.

Objective:

Primary objective

• To determine Maximum Tolerated Dose (MTD) of TH-302 combined with chemoradiotherapy (23 x 1.8 Gy in combination with Carboplatin and Paclitaxel) in patients with distal esophageal or esophago-gastric junction adenocarcinoma, and consequently find the recommended phase II dose (RP2D).

Secondary objective

* To explore the prognostic and predictive value on outcome of the repeated hypoxia PET/CT-scan at baseline and after administration of TH-302 (before start of RCT).
* To determine presence of anti-tumor activity with TH-302 administration.
* To explore the relationship between tumor hypoxia detected by the HX4 PET/CT-scans and serum biomarker expression: CAIX and Osteopontin expression.

Study design: Open-label, single-center phase 1 study of an investigational agent TH-302 and standard chemoradiotherapy with a 3+3 dose escalation design through 3 dose levels.

Number of patients: 9 to18. For each of the 3 dose steps, 3 to 6 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the esophagus
* Age >18 years
* UICC T2-4 N0-2 M0, potentially resectable disease
* Patient discussed at tumour board (multidisciplinary team meeting)
* No evident tumor invasion in nearby regions like aorta or trachea
* WHO performance status 0-2
* Less than 10 % weight loss in the past 6 months
* Laboratory requirements within 7 days prior to enrollment (start chemoradiotherapy):
* Haematology:

  * haemoglobin >10g/dl
  * absolute neutrophils ≥ 1.5 x 109/L
  * platelets ≥ 100x109/L
* Biochemistry:

  * bilirubin within institutional normal limits
  * AST(SGOT)/ALT (SGPT) ≤ 2.5 institutional upper limit
  * Creatinine clearance ≥ 60 ml/min
* Willing and able to comply with the study prescriptions
* No history of prior thoracic radiotherapy
* No severe chronic obstructive pulmonary disease with hypoxemia or in the opinion of the investigator any physiological state leading to hypoxemia
* Women should not be pregnant or lactating
* No known infection with HIV, hepatitis B or C or any other active infection
* Normal ECG with careful evaluation of QT/QTc
* Have given written informed consent before patient registration

Exclusion Criteria:

* Recent (< 3 months) severe cardiac disease (arrhythmia, congestive heart failure, infarction)
* Patients with difficult peripheral intravenous access
* History of prior thoracic radiotherapy
* severe chronic obstructive pulmonary disease with hypoxemia or in the opinion of the investigator any physiological state leading to hypoxemia
* Women who are pregnant or lactating
* Known infection with HIV, hepatitis B or C or any other active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT ) | within 30days postoperative
  To determine the DLT and define the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
hypoxia response in tumor | day 4 and day 8
  Presence of hypoxia response based on hypoxia imaging (HX4) at baseline and first administration of TH-302 (before chemoradiotherapy).
rate of pathological Complete Remission (pCR) | within 30 days after surgery
  Presence of anti-tumor activity measured by the rate of pathological Complete Remission (pCR)
histopathologic negative circumferential resection margin (CRM) rate | within 30 days after surgery
  Presence of anti-tumor activity measured by histopathologic negative circumferential resection margin (CRM) rate.
Local recurrence rate | within 30 days after surgery
  Presence of anti-tumor activity measured by local recurrence rate
distance recurrence rate | within 30 days after surgery
  Presence of anti-tumor activity measured by distance recurrence rate
Progression free survival | within 30 days after surgery
  Presence of anti-tumor activity measured by progression free survival
overall survival | within 30 days after surgery
  Presence of anti-tumor activity measured by overall survival
metabolic response | within 30 days after surgery
  Presence of anti-tumor activity measured by metabolic response one month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — MUMC+, dept Radiotherapy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larue RT, Van De Voorde L, Berbee M, van Elmpt WJ, Dubois LJ, Panth KM, Peeters SG, Claessens A, Schreurs WM, Nap M, Warmerdam FA, Erdkamp FL, Sosef MN, Lambin P. A phase 1 'window-of-opportunity' trial testing evofosfamide (TH-302), a tumour-selective hypoxia-activated cytotoxic prodrug, with preoperative chemoradiotherapy in oesophageal adenocarcinoma patients. BMC Cancer. 2016 Aug 17;16:644. doi: 10.1186/s12885-016-2709-z. PMID 27535748